CLINICAL TRIAL: NCT05830812
Title: Improving the Intraoperative Diagnosis Accuracy for Pre-invasive and Invasive Small-sized Lung Adenocarcinoma Node by Combining Multi-modal Information
Brief Title: Improving the Intraoperative Diagnosis Accuracy of Invasiveness for Small-sized Lung Adenocarcinoma
Status: Recruiting | Type: Observational
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Yang Jin, Professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Other Study IDs: HXJY20220701
Record Dates: First submitted 2023-03-24; First posted 2023-04-26 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Lung Adenocarcinoma, Stage I
Keywords: multi-modal information; lung adenocarcinoma; intraoperative diagnosis; invasiveness
MeSH Terms: conditions — Adenocarcinoma of Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- adenocarcinoma in situ: Adenocarcinoma in situ is defined as a small (≤3 cm) localized nodule with lepidic growth, mostly non-mucinous.
  Interventions: Diagnostic Test: Invasiveness diagnosis
- minimally invasive adenocarcinoma: Minimally invasive adenocarcinoma defined as a small (≤3 cm) solitary adenocarcinoma with a predominantly lepidic pattern and ≤5 mm invasion in greatest dimension.
  Interventions: Diagnostic Test: Invasiveness diagnosis
- invasive adenocarcinoma: Invasive adenocarcinoma is a malignant epithelial tumor with glandular differentiation, mucin production, or pneumocyte marker expression. The tumors show an acinar, papillary, micropapillary, lepidic, or solid growth pattern, with either mucin or pneumocyte marker expression. The invasive ademocarcinoma component should be present in at least one focus measuring >5mm in greatest dimension.
  Interventions: Diagnostic Test: Invasiveness diagnosis

INTERVENTIONS:
Diagnostic Test: Invasiveness diagnosis — To predict the invasiveness of patients with small-sized lung adenocarcinoma intraoperatively based on multi-modal information.

SUMMARY:
The goal of this observational study is to improve the intraoperative diagnosis accuracy of invasiveness for small-sized lung adenocarcinoma by combining multi-modal information. The main question it aims to answer is whether multi-modal information have great value of prediction on the invasiveness for small-sized lung adenocarcinoma. Since a promising limited resection is largely based on intraoperative frozen section diagnosis, there is a growing demand on the high-accuracy of timely pathology diagnosis. The multi-modal information of participants will be collected retrospectively.

ELIGIBILITY:
Inclusion Criteria:

CT examination within 3 months before surgery Patients with operable clinical stage I lung cancer No previous treatment in the lungs or any other organ

≥ 20 years and ≤ 80 years old Tumor less than 3cm in diameter on thin-slice (0.625-1 mm) CT images Lung adenocarcinoma confirmed by surgical resection and histopathological diagnosis

Exclusion Criteria:

Marked artifacts on CT images History of preoperative treatment Incomplete clinical information or DICOM images History of other malignant tumors Lung cancer associated with cystic airspaces

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From January 2018 to December 2022, about 3000 patients with lung adenocarcinoma were enrolled in this retrospective study.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Final pathology diagnosis of the paraffin section stained with HE | Immediately after operation
  The final pathology diagnosis after resection

CONTACTS AND LOCATIONS:
Overall Officials: Yang Jin, PHD, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No